CLINICAL TRIAL: NCT00233103
Title: Treatment of Post-TBI Depression
Brief Title: Treatment of Post-Traumatic Brain Injury (TBI) Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 02-0677; H133A020501
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Results first posted 2015-11-13 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-10

CONDITIONS: Depression
Keywords: Sertraline; TBI; depression; SSRI; brain injury
MeSH Terms: conditions — Depression; Brain Injuries | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sertraline (Experimental): Daily oral sertraline in doses starting at 25mg and increasing to therapeutic levels (up to 200mg).
  Interventions: Drug: Sertraline
- Placebo (Placebo Comparator): Placebo for 10 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sertraline — Sertraline arm
  Arms: Sertraline
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Randomized clinical trial of sertraline vs. placebo for post-TBI depression

DETAILED DESCRIPTION:
Purpose: The purpose of this study is to document the efficacy of sertraline (Zoloft) in the treatment of depression (major depressive disorder) after TBI, including the impact on quality of life. Researchers will also explore the effects of sertraline on anxiety disorders, which often accompany post-TBI depression.

Background: Major depression is experienced by many more people after TBI than prior to injury and more often than in people without a brain injury. Many studies have also shown that this higher than 'normal' incidence looms for many years post TBI. Major depression is associated with a variety of negative outcomes, including poorer functioning in basic activities, reduced employment, elevated divorce rate, reduced social and recreational activity and increased sexual dysfunction.

Need for Research: Of the current drug treatments for major depression, sertraline and similar drugs (known as selective serotonin reuptake inhibitors, or selective serotonin reuptake inhibitor (SSRIs)) have few side effects in people who have experienced a brain injury and have been shown to be effective in people with no known brain injury. However, information on the impact of SSRIs on post-TBI depression, based on randomized, double-blind studies, is unavailable.

Current Research Activity: Approximately 50 men and women volunteers who are post TBI and currently diagnosed with major depressive disorder are being randomly assigned to a 12-week period of taking Zoloft or a placebo. Over the period of study, participants will have the severity of their depressive symptoms assessed (as well as their symptoms of anxiety); a simple measure of the volunteer's perceived quality of life will be implemented prior to the study and at its termination. It is hypothesized that sertraline will reduce the symptoms of depression and anxiety and will increase the person's perceived quality of life to a significantly greater extent than will the placebo.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* experienced a TBI with a documented loss of consciousness or other evidence of a TBI (i.e., evidence of pathology on neuro-imaging)
* at least 6 months post-injury
* English-speaking
* residential telephone service
* living within 1.5 hours of New York City
* able to comprehend or answer verbal or written questionnaires
* willing to provide consent to participate in a 12 week drug study to treat Major Depressive Disorder (MDD); current MDD as diagnosed using Structured Clinical Interview for Diagnostic and Statistical Manual Diploma in Social Medicine (DSM) Disorders (SCID), and severity of MDD rated at least 18 on the HAM-D.

Exclusion Criteria:

* currently taking antidepressant medication (including monamine oxidase inhibitors (MOAs) or tricyclic antidepressants (TCAs)
* unwilling to abstain from seeking new psychosocial or pharmacologic treatments during the course of the study
* currently in psychotherapy
* active suicidal plans and/or requiring hospitalization
* prior use of sertraline
* currently experiencing other serious medical illness
* currently pregnant or breast feeding
* mass brain lesions or other neurological diagnoses other than TBI
* history of current or past psychosis or mania
* current substance abuse
* history of clinically significant liver or renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2003-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Gordon, Ph.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Ashman TA, Cantor JB, Gordon WA, Spielman L, Flanagan S, Ginsberg A, Engmann C, Egan M, Ambrose F, Greenwald B. A randomized controlled trial of sertraline for the treatment of depression in persons with traumatic brain injury. Arch Phys Med Rehabil. 2009 May;90(5):733-40. doi: 10.1016/j.apmr.2008.11.005. PMID 19406291

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through physician referrals and flyers posted in outpatient rehabilitation treatment areas and distributed at TBI-survivor groups. Participants from past research projects who had agreed to be contacted for future studies were contacted.
Groups:
- Sertraline: Daily oral sertraline in doses starting at 25mg and increasing to therapeutic levels (up to 200mg) for 10 weeks
Period: Overall Study
Arm/Group | Sertraline | Placebo
Started | 27 | 25
Completed | 22 | 19
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sertraline | Placebo | Total
Number analyzed (Participants) | 22 | 19 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (12.8) | 51.5 (8.2) | 49.1 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 19
  Male | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Depression at Baseline
Description: The 17-item Hamilton Rating Scale for Depression (HAM-D) is a widely used clinician-rated measurement of depression severity. A score of 0-7 is considered to be normal. 8-13 = mild depression, 14-18 = moderate depression, 19-22 = severe depression, and ≥ 23 = very severe depression.
  Self-report of depression and DSM-IV diagnosis (HAM-D score) at baseline.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 22 | 19
units on a scale | 27.5 (7.1) | 25.2 (8.0)

2. Secondary Outcome: BAI
Description: The Beck Anxiety Inventory (BAI) is a 21-item self-report measure that assesses subjective, somatic, or panic-related symptoms associated with anxiety rated on a scale from 0 (not at all) to 3(severely). Total score: 0-7 = minimal level of anxiety, 8-15 = mild anxiety, 16-25 = moderate anxiety, and 26-63 = severe depression
Time Frame: Immediately post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 22 | 19
units on a scale | 11.1 (11.9) | 13.1 (11.6)

3. Secondary Outcome: Life-3
Description: Life-3 is a single-item Quality of life (QOL) measure that uses a 7-point Likert-type scale to assess satisfaction with life during the past month. It is typically administered twice during an evaluation, and the mean of the 2 obtained scores is used. Higher scores on this measure indicate higher levels of subjective QOL. Range from 1 to 7.
Time Frame: Immediately post-intervention at 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 22 | 19
units on a scale | 6.3 (8.0) | 4.9 (3.5)

4. Primary Outcome: Depression at End of Treatment
Description: Self-report of depression and Diagnostic and Statistical Manual Diploma in Social Medicine (DSM-IV) diagnosis (HAM-D score) compared at end of treatment to baseline. Participants were considered treatment responders if their initial HAM-D decreased by 50% or dropped below a score of 10 at the end of the intervention.
  The 17-item Hamilton Rating Scale for Depression (HAM-D) is a widely used clinician-rated measurement of depression severity. A score of 0-7 is considered to be normal. 8-13 = mild depression, 14-18 = moderate depression, 19-22 = severe depression, and ≥ 23 = very severe depression.
Time Frame: end of treatment, average of 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 22 | 19
units on a scale | 13.7 (9.7) | 16.2 (9.6)

ADVERSE EVENTS:
Arm/Group | Sertraline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/19
Other Adverse Events (participants affected / at risk) | 1/22 | 2/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline (N=22) | Placebo (N=19)
anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
depression (Psychiatric disorders) | 0 (0) | 1 (1)
allergic reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Sample size was small - those who dropped out could have reduced the differential effect.

Sample was heterogeneous for severity and time since injury.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes